CLINICAL TRIAL: NCT01160991
Title: Effects of the Serotonin 2A Receptor on Insulin Sensitivity and Secretion: a Double-blind Controlled Comparison of Olanzapine vs. Amisulpride:
Brief Title: Effect of Atypical Antipsychotic Drugs Olanzapine and Amisulpride on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Michael Deuschle, Central Institute of Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DeuOlanAmi
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenia; Diabetes; Insulin Resistance
Keywords: schizophrenia; olanzapine; atypical antipsychotic drugs; amisulpride; diabetes; insulin resistance; insulin secretion; glucose; euglycemic hyperinsulinemic clamp; hyperglycemic clamp
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Insulin Resistance | interventions — Glucose Clamp Technique; Amisulpride; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amisulpride (Active Comparator): Single dose of amisulpride 200 mg p.o. given at 8:00 a.m.
  Interventions: Procedure: Glucose clamp technique; Drug: Amisulpride
- Olanzapine (Experimental): Single dose of olanzapine 10 mg p.o. given at 8:00 a.m.
  Interventions: Procedure: Glucose clamp technique; Drug: Olanzapine
- Placebo (Placebo Comparator): Placebo capsules are given at 8:00 a.m. Procedures are performed as described above.
  Interventions: Procedure: Glucose clamp technique; Drug: Placebo

INTERVENTIONS:
Procedure: Glucose clamp technique — euglycemic hyperinsulinemic clamp with target blood glucose of 90 mg/dl (5 mmol/l), followed by hyperglycemic clamp, target blood glucose of 180 mg/dl (10 mmol/l) for measurement of insulin sensitivity and insulin secretion
Drug: Amisulpride — Single dose of amisulpride 200 mg p.o. given at 8:00 a.m.
  Arms: Amisulpride
Drug: Olanzapine — Single dose of olanzapine 10 mg p.o. given at 8:00 a.m.
  Arms: Olanzapine
Drug: Placebo — Placebo capsules are given at 8:00 a.m.
  Arms: Placebo

SUMMARY:
Patients suffering from schizophrenia have a high risk to become obese and develop diabetes. Risk of obesity is particularly high with some newer schizophrenia drugs, such as clozapine or olanzapine. These drugs are called atypical drugs and exert their action in part by occupying receptors for serotonin, particularly the 5HT2A receptor subtype. This receptor may also interfere with glucose metabolism and insulin action. The purpose of this study is to compare an atypical antipsychotic drugs, olanzapine, which acts by occupying the 5HT2A receptor, to another antipsychotic drug, amisulpride, which mainly acts through the dopamine pathway. Healthy volunteers are recruited and asked to take a single dose of each drug and of placebo on separate days. Then, a combined glucose clamp study will be performed in order to test the effects of these drugs on insulin sensitivity and insulin secretion.

DETAILED DESCRIPTION:
10 male healthy volunteers are recruited. After informed consent, they are admitted to the study ward at 10:00 p.m. prior to the study day and kept fasting until the next morning. At 8:00 a.m. they receive their study medication (olanzapine, amisulpride or placebo). Subsequently, measurements of insulin sensitivity and insulin secretion are performed by euglycemic hyperinsulinemic clamp technique followed by hyperglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers
* written informed consent

Exclusion Criteria:

* BMI > 30 kg/m²
* Diabetes mellitus
* Hypertension
* Treatment with drugs interfering with lipid or glucose metabolism (e.g. statins, oral antidiabetic drugs, glucocorticoids)
* History of seizures

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 90 thru 120 min after application of study drug
  m-value during euglycemic glucose clamp (glucose infusion rate divided by time and body weight)

SECONDARY OUTCOMES:
pancratic c-peptide secretion | 120 thru 180 minutes after administration of study drug
  C-peptide measured 4 times during hyperglycemic clamp period at time 0 min (prior to glucose bolus), 5 min, 10 min and 60 min after glucose bolus

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kopf, M.D., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany